CLINICAL TRIAL: NCT02462083
Title: A Phase 3, Multicenter, Open Label Study to Evaluate the Long-Term Safety of IDP-118 Lotion in the Treatment of Plaque Psoriasis
Brief Title: Long-Term Safety of IDP-118 Lotion in the Treatment of Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Dow Pharmaceutical Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V01-118A-303; NCT02611349 (obsolete NCT alias)
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Results first posted 2020-01-27 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IDP-118 Lotion (Experimental): IDP-118 lotion (halobetasol propionate 0.01%, tazarotene 0.045%) will be applied topically on the affected area once daily for 8 weeks and then as needed once daily for up to 1 year.
  Interventions: Drug: IDP-118 Lotion

INTERVENTIONS:
Drug: IDP-118 Lotion — IDP-118 lotion will be applied as per the instructions provided by the investigational center staff.

SUMMARY:
The objective of this study is to evaluate the long-term safety of IDP-118 lotion.

DETAILED DESCRIPTION:
This is a multicenter, open-label study of the long-term safety of IDP-118 lotion in participants with plaque psoriasis.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female, of any race, at least 18 years of age (inclusive).
* Freely provides both verbal and written informed consent.
* Has an area of plaque psoriasis appropriate for topical treatment that covers a Body Surface Area (BSA) of at least 3 percent (%), but no more than 12%. The face, scalp, palms, soles, axillae and intertriginous areas are to be excluded in this calculation.
* Is willing and able to avoid prolonged exposure of the treatment area to ultraviolet radiation (natural and artificial) for the duration of the study.
* Has a clinical diagnosis of psoriasis at the Baseline visit with an Investigators Global Assessment (IGA) score of 3 or 4 (The face, scalp, palms, soles, axillae and intertriginous areas are to be excluded in this assessment).

Key Exclusion Criteria:

* Has spontaneously improving or rapidly deteriorating plaque psoriasis or pustular psoriasis, as determined by the investigator.
* Presents with psoriasis that was treated with prescription medication and failed to respond to treatment, even partially or temporarily, as determined by the Investigator.
* Presents with any concurrent skin condition that could interfere with the evaluation of the treatment areas, as determined by the investigator.
* Is pregnant, nursing an infant, or planning a pregnancy during the study period.
* Has received treatment with any investigational drug or device within 60 days or 5 drug half lives (whichever is longer) prior to the Baseline visit, or is concurrently participating in another clinical study with an investigational drug or device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2015-08-11 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Binu J Alexander, Study Director — Valeant Pharmaceuticals
Locations (46):
- United States (46):
  - Valeant Site 6, Mobile, Alabama
  - Valeant Site 24, Beverly Hills, California
  - Valeant Site 32, Encinitas, California
  - Valeant Site 27, Encino, California
  - Valeant Site 33, Los Angeles, California
  - Valeant Site 43, Los Angeles, California
  - Valeant Site 45, Sacramento, California
  - Valeant Site 25, San Diego, California
  - Valeant Site 4, San Diego, California
  - Valeant Site 44, Santa Monica, California
  - Valeant Site 36, Santa Rosa, California
  - Valeant Site 10, Englewood, Colorado
  - Valeant Site 3, Boynton Beach, Florida
  - Valeant Site 28, Coral Gables, Florida
  - Valeant Site 1, Miami, Florida
  - Valeant Site 37, North Miami Beach, Florida
  - Valeant Site 13, Sanford, Florida
  - Valeant Site 41, Snellville, Georgia
  - Valeant Site 17, South Bend, Indiana
  - Valeant Site 12, Olathe, Kansas
  - Valeant Site 19, Louisville, Kentucky
  - Valeant Site 14, Louisville, Kentucky
  - Valeant Site 35, Clinton Township, Michigan
  - Valeant Site 34, Detroit, Michigan
  - Valeant Site 16, Warren, Michigan
  - Valeant Site 18, Fridley, Minnesota
  - Valeant Site 31, Omaha, Nebraska
  - Valeant Site 2, East Windsor, New Jersey
  - Valeant Site 29, New York, New York
  - Valeant Site 39, Rochester, New York
  - Valeant Site 5, Portland, Oregon
  - Valeant Site 11, Philadelphia, Pennsylvania
  - Valeant Site 30, Charleston, South Carolina
  - Valeant Site 15, Nashville, Tennessee
  - Valeant Site 9, Dallas, Texas
  - Valeant Site 40, Houston, Texas
  - Valeant Site 8, Houston, Texas
  - Valeant Site 46, Katy, Texas
  - Valeant Site 20, Pflugerville, Texas
  - Valeant Site 21, San Antonio, Texas
  - Valeant Site 7, San Antonio, Texas
  - Valeant Site 22, Webster, Texas
  - Valeant Site 38, Salt Lake City, Utah
  - Valeant Site 23, Lynchburg, Virginia
  - Valeant Site 26, Norfolk, Virginia
  - Valeant Site 42, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- IDP-18 Lotion: IDP-118 Lotion (HP 0.01%, Taz 0.045%) was applied topically on the affected area once daily for 8 weeks and then as needed once daily for up to 1 year.
Period: Overall Study
Arm/Group | IDP-18 Lotion
Started | 555
Safety Population (All participants with >=1 confirmed dose of study drug & >=1 post-Baseline safety assessment.) | 550
Completed | 136
Not Completed | 419
Not completed — Sponsor request | 39
Not completed — Withdrawal by Subject | 87
Not completed — Lost to Follow-up | 41
Not completed — Lack of Efficacy | 151
Not completed — Pregnancy | 1
Not completed — Protocol Violation | 6
Not completed — Adverse Event | 33
Not completed — Worsening condition | 16
Not completed — Other than specified | 45

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one confirmed dose of study drug and had at least one post-baseline safety assessment.
Groups:
- IDP-118 Lotion: IDP-118 Lotion (HP 0.01%, Taz 0.045%) was applied topically on the affected area once daily for 8 weeks and then as needed once daily for up to 1 year.
Arm/Group | IDP-118 Lotion
Number analyzed (Participants) | 550
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (14.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 189
  Male | 361
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 141
  Not Hispanic or Latino | 409
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 15
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 46
  White | 473
  More than one race | 0
  Unknown or Not Reported | 12

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Grade 3 Local Skin Reactions
Description: Local skin reactions (itching, dryness, burning/stinging) graded at a level of 3 (severe) at any point in the study following the first application of study drug were assessed. Severe Itching (as reported by the participant within the last 24 hours) referred to the intense itching that may interrupt daily activities and/or sleep. Severe dryness (as assessed by the investigator) referred to as marked roughness of the skin. Severe burning/stinging (as reported by the participant within the last 24 hours) referred to as hot burning sensation that causes definite discomfort and may interrupt daily activities and/or sleep. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Baseline up to Week 52
Population: as for baseline characteristics
Measure: Number; unit: percentage of participants
Arm/Group | IDP-118 Lotion
Number analyzed (Participants) | 550
percentage of participants
  Itching | 22.2
  Dryness | 6.9
  Burning/stinging | 9.8

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: Safety population included all participants who received at least one confirmed dose of study drug and had at least one post-baseline safety assessment.
Arm/Group | IDP-118 Lotion
All-Cause Mortality (participants affected / at risk) | 0/550
Serious Adverse Events (participants affected / at risk) | 18/550
Other Adverse Events (participants affected / at risk) | 131/550
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-118 Lotion (N=550)
Cellulitis gangrenous (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Colitis ulcerative (Gastrointestinal disorders) | 1
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Small intestine adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Intervertebral disc operation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IDP-118 Lotion (N=550)
Application site dermatitis (General disorders) | 59
Application site pruritus (General disorders) | 33
Application site pain (General disorders) | 29
Nasopharyngitis (Infections and infestations) | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT02462083/Prot_SAP_000.pdf